CLINICAL TRIAL: NCT01352728
Title: A Phase II Study of Transarterial Chemoembolisation and Axitinib for the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Hepatocellular Carcinoma (HCC) Transarterial Chemoembolisation (TACE) +Axitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC028
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TACE+Axitinib (Experimental)
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — 5 mg daily for 6 cycle with TACE+Axitinib, Axitinib continued until PD.

SUMMARY:
The survival of subjects with unresectable hepatocellular carcinoma (HCC) receiving transarterial chemoembolization is improved with addition of axitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HCC (or fulfilling AASLD criteria for HCC diagnosis in HBsAg positive subjects with cirrhosis in case biopsy is not feasible)
2. Disease must not be amenable to potentially curative surgery
3. Without prior systemic nor transarterial treatment
4. Prior surgery or local therapy is allowed but the target lesion must have not been previously treated
5. Child-Pugh stage A liver function
6. ECOG performance 0-2
7. Life expectancy longer than 12 weeks
8. At least one measurable treatment lesion according to modified RECIST criteria
9. Adequate haematological, hepatic and renal function

Exclusion Criteria:

1. Contra-indications to TACE treatment:

   * Main portal vein thrombosis or occlusion
   * Evidence of biliary obstruction
   * Presence of extra-hepatic disease
2. Diffuse-type HCC
3. Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment.
4. Any form of prior transarterial therapy or systemic therapy for HCC.
5. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors or CYP3A4 or CYP1A2 inducers.
6. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
7. Any haemorrhage or bleeding event of CTCAE Grade 3 or more within 4 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05-18 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Two-year survival rate | 4 years

SECONDARY OUTCOMES:
Overall confirmed objective response rate (ORR) as determined according to modified RECIST. | 4 years
Disease Control Rate (DCR) | 4 Years
Duration of Response (DR) | 4 years
Time to Progression (TTP) | 4 years
Progression-Free Survival (PFS) | 4 years
Overall survival (OS) | 4 years
Type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities | 4 years
Quality of Life | 4 years
Tissue and Serum Biomarkers | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Chan, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan SL, Yeo W, Mo F, Chan AWH, Koh J, Li L, Hui EP, Chong CCN, Lai PBS, Mok TSK, Yu SCH. A phase 2 study of the efficacy and biomarker on the combination of transarterial chemoembolization and axitinib in the treatment of inoperable hepatocellular carcinoma. Cancer. 2017 Oct 15;123(20):3977-3985. doi: 10.1002/cncr.30825. Epub 2017 Jun 22. PMID 28640364